CLINICAL TRIAL: NCT05533099
Title: A Pilot Study of REGENERA Implant in Localized Non-malignant Breast Lesions Treated by Excision or Lumpectomy - Long-term Follow-up
Brief Title: REGENERA Implant in Localized Non-malignant Breast Lesions Treated by Excision or Lumpectomy - Long-term Follow-up
Status: Active, not recruiting | Type: Observational
Sponsor: Tensive SRL (Industry)
Collaborators: Advice Pharma Group srl (Industry)
Responsible Party: Sponsor
Other Study IDs: Tens-BBC/002/2020
Record Dates: First submitted 2022-09-06; First posted 2022-09-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Breast Diseases
MeSH Terms: conditions — Breast Diseases | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — Observational study of a device implanted in a previous clinical study

SUMMARY:
In a previous first-in-human (FIH) study we assessed safety and performance of REGENERA in 15 patients treated for breast deformities following excision or lumpectomy. The technique was minimally invasive, easily repeated and associated with minimal surgical morbidity.

It is important to assess whether the positive safety and performance results obtained during the initial 6 months post- surgery are maintained in the long-term, for up to 5 years after surgery.

In this long-term follow-up study we will assess long-term safety and performance of REGENERA implant after excision or lumpectomy of breast tissue in patients with non-malignant lesions.

DETAILED DESCRIPTION:
REGENERA is a polymeric bioresorbable scaffold. The REGENERA matrix is characterized by an interconnected open pore/void structure, having average pore/void diameter from 0.3 to 6.5 mm and local thickness of 30 μm ± 20 μm (μCT 50, SCANCO Medical AG, Brüttisellen, Switzerland). A network of channels is embedded into the porous structure according to a specific pattern, where the channels are interconnected with the porous structure.

The biomaterial constituting REGENERA is composed of a patented biodegradable cross-linked poly(urethane-ester- ether) foam coated with a bio adhesive macromolecule [Poly(L- lysine); PLL] and hydrophobized by Oleic acid (18:1 n-9), a monounsaturated fatty acid.

The shape and geometry of REGENERA have been set to facilitate its insertion to the implantation site and to fulfill the volume deficit caused by excision of lesioned soft tissue after lumpectomy.

REGENERA is a polymeric bioresorbable scaffold intended to support the ingrowth of the patient's soft tissue when used to restore the natural appearance of the breast after surgical removal of benign and malignant breast lesions, up to 200 cc in volume.

In this long-term follow-up study we will assess long-term safety and performance of REGENERA implant after excision or lumpectomy of breast tissue in patients with non-malignant lesions.

REGENERA is the first medical device designed to restore a natural breast, after breast-conserving surgery (lumpectomy). As shown by the preliminary results of the FIH pilot study, a natural shape and feeling could be achieved, based on the patient's soft tissue growth ability, in a single step, easy-to- adopt and, potentially, cost saving procedure, for the healthcare stakeholders. The few post-operative complications combined with the positive psychological impact generated by the existence of a valid reconstructive option after lumpectomy, has the potential to improve the patients' quality of life, during and after post-surgery recovery.

Because all of that, the purpose of this long-term follow-up study is to assess whether REGENERA does not cause long-term safety issues and confirms its performance in the long-term.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with REGENERA according to protocol Tens-BBC/001/2017
* Patients able and willing to give written informed consent form

Exclusion Criteria:

- There are no formal exclusion criteria for participation, as this LTFU study aims at following all the patients who have completed protocol Tens-BBC/001/2017, subject to informed consent.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female adult subjects diagnosed with localized, non-malignant breast lesions, who underwent surgery with REGENERA implant after excision or lumpectomy of breast tissue, according to protocol Tens-BBC/001/2017
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2026-05-17 (Estimated); Study Completion 2026-05-17 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events | 54 months
  Rate of adverse events associated with the device (REGENERA implant)

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Roncella, MD, Principal Investigator — Unità Operativa di Senologia (Breast Surgery Unit), Ospedale Santa Chiara
Locations (1):
- Unità Operativa di Senologia (Breast Surgery Unit), Ospedale Santa Chiara, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mariniello MD, Roncella M, Mazzotta D, Gerges I, Colizzi L, Tamplenizza M, Tocchio A, Martello F, Ghilardi M, Cossu MC, Danti S, Ghilli M. Scaffold-based breast conserving surgery in patients with non-malignant breast lesions: long-term follow-up of a first-in-human pilot study on the REGENERA biomimetic breast implant. Breast Cancer. 2026 Jan;33(1):111-122. doi: 10.1007/s12282-025-01780-w. Epub 2025 Sep 27. PMID 41014462